CLINICAL TRIAL: NCT04392037
Title: A Phase 2 Study of CC220 (Iberdomide) Combined With Low-dose Cyclophosphamide and Dexamethasone in Relapsed/Refractory Multiple Myeloma (IberCd): ICON Study
Brief Title: Iberdomide Combined With Low-dose Cyclophosphamide and Dexamethasone
Acronym: ICON
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Amsterdam UMC, location VUmc (Other)
Collaborators: Celgene (Industry)
Responsible Party: Principal Investigator, WCJ van de Donk, Prof. Niels W.C.J. van de Donk, Amsterdam UMC, location VUmc
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HAEM-2020-1; NL72835.029.20 (Other: Toetsing Online); 2019-004604-35 (EudraCT Number)
Record Dates: First submitted 2020-05-13; First posted 2020-05-18 (Actual); Last update posted 2025-03-28 (Actual); Status verified 2025-03

CONDITIONS: Multiple Myeloma
MeSH Terms: conditions — Multiple Myeloma | interventions — iberdomide; Cyclophosphamide; Dexamethasone

STUDY DESIGN:
Intervention Model Description: Patients will be treated with iberdomide plus low-dose cyclophosphamide and dexamethasone (IberCd)
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- Iberdomide plus low-dose cyclophosphamide and dexamethasone (Experimental): Iberdomide 1.6mg on days 1-21
  Low-dose Cyclophosphamide 50 mg on days 1-28 of each 28 day cycle
  Dexamethasone 40 mg once weekly (20 mg in patients aged > 75 years)
  Interventions: Drug: Iberdomide plus low-dose cyclophosphamide and dexamethasone

INTERVENTIONS:
Drug: Iberdomide plus low-dose cyclophosphamide and dexamethasone — Iberdomide, low dose Cyclophosphamide and Dexamethason will be given until progression or unacceptable toxicity
  Other Names: CC-220

SUMMARY:
Evaluation of the effect iberdomide combined with low-dose cyclophosphamide and dexamethasone in patients with relapsed/refractory multiple myeloma.

DETAILED DESCRIPTION:
Novel drugs such as lenalidomide (an immunomodulatory drug; IMiD) have markedly improved the prognosis of multiple myeloma patients. Over the recent years, lenalidomide is increasingly used as part of first line therapy, typically until the development of progressive disease. These lenalidomide-refractory patients can be treated with several regimens. However, these regimens frequently contain proteasome inhibitors which are associated with neuropathy (bortezomib) or cardiovascular complications (carfilzomib). These proteasome inhibitors also need to be administered subcutaneously or intravenously in the hospital, once or twice per week. Also these regimens have limited efficacy in lenalidomide-refractory patients. This indicates that there is still an unmet medical need for new treatment options for patients who develop lenalidomide-refractory disease. These new treatment regimens should be active and safe without induction of neuropathy or cardiovascular side effects Moreover, an all oral regimen is frequently preferred by patients.

Iberdomide plus low-dose cyclophosphamide and dexamethasone

Available data indicates that the Cereblon E3 ligase modifying drug (CELMoD) iberdomide (CC220) is pharmacologically distinct from lenalidomide and pomalidomide with a higher potency against Cereblon, leading to differentiated antitumor and immunostimulating effects. Since iberdomide plus dexamethasone is active and well-tolerated in heavily pretreated patients including those with lenalidomide/pomalidomide-refractory disease, this two-drug regimen forms a new platform to which other agents can be added. The combinations of bortezomib, carfilzomib, or daratumumab plus iberdomide and dexamethasone are currently being evaluated.

Investigators have shown that low-dose cyclophosphamide can be effectively combined with the IMiDs lenalidomide and pomalidomide. These combinations are effective and are well-tolerated.

To address the unmet medical need for new treatment options for lenalidomide-refractory MM patients, the investigators aim at further improving the efficacy of IMiD/CELMoD plus dexamethasone combination therapy in terms of response and progression-free survival, by adding low-dose cyclophosphamide to the iberdomide-dexamethasone backbone (IberCd). This all-oral regimen will be tested in a lenalidomide-refractory patient population with 2-4 prior lines of therapy. The goal of this trial is to investigate the efficacy and safety of the IberCd combination in multiple myeloma patients who have refractory disease or a relapse after prior treatment with lenalidomide. Besides, various correlative studies will be performed during this trial including immune monitoring.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Subject must have documented diagnosis of multiple myeloma and have measurable disease as defined by any of the following:

   • Serum monoclonal paraprotein (M-protein) level ≥5 g/L (0.5 g/dL); or urine M-protein level ≥200 mg/24 hours; or serum immunoglobulin free light chain ≥100 mg/L (10 mg/dL) and abnormal serum immunoglobulin kappa lambda free light chain ratio (See Appendix A)
3. Relapsed or refractory disease. Relapse is defined as progression of disease after an initial response to previous treatment, more than 60 days after cessation of treatment. Refractory disease is defined as <50% reduction in M-protein or progression of disease during treatment or within 60 days after cessation of treatment.
4. Subject had 2-4 prior anti-myeloma regimens. (Note: Induction, bone marrow transplant with or without maintenance therapy is considered one regimen; Prior pomalidomide is allowed )
5. Subject has developed lenalidomide-refractory disease (any dose) during prior treatment with lenalidomide or a lenalidomide-containing regimen Lenalidomide-refractory MM is defined as progressive disease during therapy, no response (< PR) to prior lenalidomide-containing therapy, or progression within 60 days of discontinuation from lenalidomide-containing regimens, according to the International Myeloma Working Group criteria.
6. WHO performance 0, 1, or 2
7. Life expectancy at least 3 months
8. Written informed consent
9. A female of childbearing potential (FCBP) is a female who: 1) has achieved menarche at some point, 2) has not undergone a hysterectomy or bilateral oophorectomy, or 3) has not been naturally postmenopausal (amenorrhea following cancer therapy does not rule out childbearing potential) for at least 24 consecutive months (i.e., has had menses at any time in the preceding 24 consecutive months) and must:

   1. Have two negative pregnancy tests as verified by the Investigator prior to starting study treatment. She must agree to ongoing pregnancy testing during the course of the study, and after end of study treatment. This applies even if the subject practices true abstinence* from heterosexual contact.
   2. Either commit to true abstinence* from heterosexual contact (which must be reviewed on a monthly basis and source documented) or agree to use, and be able to comply with two forms of contraception: one highly effective, and one additional effective (barrier) measure of contraception without interruption 28 days prior to starting investigational product, during the study treatment (including dose interruptions), and for at least 28 days after the last dose of CC-220, 90 days after the last dose of cyclophosphamide, whichever is longer. Contraception requirements are detailed in Appendix H.
10. Male subjects must:

    a. Practice true abstinence* (which must be reviewed on a monthly basis and source documented) or agree to use a condom during sexual contact with a pregnant female or a female of childbearing potential while participating in the study, during dose interruptions and for at least 90 days following the last dose of study treatment, even if he has undergone a successful vasectomy.

    * True abstinence is acceptable when this is in line with the preferred and usual lifestyle of the subject. [Periodic abstinence (eg, calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.]
11. Males must agree to refrain from donating sperm while on study treatment, during dose interruptions and for at least 90 days following last dose of study treatment.
12. All subjects must agree to refrain from donating blood while on study treatment, during dose interruptions and for at least 28 days following the last dose of study treatment.
13. All male and female subjects must follow all requirements defined in the Pregnancy Prevention Program (v5.1). See Appendix H for CC-220 Pregnancy Prevention Plan for Subjects in Clinical Trials.

Exclusion Criteria:

1. Subjects who previously received continuous low-dose cyclophosphamide alone or in combination with other anti-MM agents are excluded (cyclophosphamide once weekly such as in bortezomib-cyclophospahmide-dexametahsone regimen (VCD) is allowed).
2. Treatment with prior iberdomide
3. Non-secretory MM
4. Systemic AL amyloidosis or plasma cell leukemia (>2.0x109/L circulating plasma cells by standard differential) or Waldenstrom's macroglobulinemia
5. Subject has known meningeal involvement of multiple myeloma
6. Inadequate marrow reserve as defined by a platelet count <75 x 109/L or an absolute neutrophil count <1.0 x 109/L
7. Corrected serum calcium >13.5 mg/dL (>3.4 mmol/L)
8. Subject has a history of anaphylaxis or hypersensitivity to thalidomide, lenalidomide, pomalidomide, dexamethasone, or cyclophosphamide. Subject has known or suspected hypersensitivity to the excipients contained in the formulation of iberdomide, dexamethasone, or cyclophosphamide.
9. Subject has received any of the following within the last 14 days of initiating IberCd:

   * Plasmapheresis
   * Major surgery (as defined by the Investigator)
   * Radiation therapy other than local therapy for MM associated bone lesions
   * Use of any systemic myeloma drug therapy
10. Subject has been treated with an investigational agent (ie, an agent not commercially available) within 28 days or 5 half-lives (whichever is longer) of initiating IberCd treatment
11. Subject has current or prior use of immunosuppressive medication within 14 days prior to the first dose of IP. The following are exceptions to this criterion:

    * Intranasal, inhaled, topical or local steroid injections (eg, intra-articular injection)
    * Systemic corticosteroids at physiologic doses that do not exceed 10 mg/day of prednisone or equivalent
    * Steroids as premedication for hypersensitivity reactions (eg, computed tomography [CT] scan premedication)
12. Subject has taken a strong inhibitor or inducer of CYP3A4/5 including grapefruit, St.

    John's Wort or related products within two weeks prior to dosing and during the course of study
13. Creatinine clearance <30 ml/min or requirement of dialysis.
14. Uncontrolled or severe cardiovascular disease (NYHA class III or IV heart failure; myocardial infarction within the last 6 months of study entry); unstable angina; unstable cardiac arrhythmias; clinically significant pericardial disease)
15. Significant hepatic dysfunction (total bilirubin ≥ 3 times normal value or transaminases ≥ 3 times normal value), unless related to myeloma
16. Subject has any concurrent severe and/or uncontrolled medical condition (e.g. uncontrolled diabetes, respiratory disease, infection, hypertension, etc.) that is likely to interfere with study procedures or results, or that in the opinion of the investigator would constitute a hazard for participating in this study.
17. Subject known to test positive for human immunodeficiency virus (HIV), chronic or active hepatitis B, or active hepatitis A or C
18. Peripheral neuropathy of ≥grade 2.
19. Subjects with gastrointestinal disease that may significantly alter the absorption of CC-220
20. History of active malignancy during the past 3 years, except squamous cell and basal cell carcinomas of the skin and carcinoma in situ of the cervix or breast and incidental histologic finding of prostate cancer (T1a or T1b using the TNM [tumor, nodes, metastasis] clinical staging system) or prostate cancer that is cured, or malignancy that in the opinion of the local investigator, with concurrence with the principal investigator, is considered cured with minimal risk of recurrence within 3 years.
21. Subject is known or suspected of not being able to comply with the study protocol (eg, because of alcoholism, drug dependency, or psychological disorder) or the subject has any condition for which, in the opinion of the investigator, participation would not be in the best interest of the subject (eg, compromise their well-being) or that could prevent, limit, or confound the protocol-specified assessments.
22. Subject is a female who is pregnant, nursing or breastfeeding, or who intends to become pregnant during the participation in the study
23. Subject is unable or unwilling to undergo protocol required thromboembolism prophylaxis
24. Subject has previously received an allogeneic stem cell transplantation within 1 year before the date of registration and has not used immunosuppressive drugs within one month before the date of registration.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2021-02-17 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Progression free survival | up to 5 years
  PFS; i.e. time from the first dose of iberdomide-cyclophosphamide-dexamethasone to progression or death from any cause, whichever comes first

SECONDARY OUTCOMES:
Overall response rate | up to 5 years
  In this analysis the investigators will consider the best response obtained during treatment according to the international myeloma working group (IMWG) criteria
Safety and toxicity | up to 5 years
  defined by type, frequency and severity of adverse events as defined by the National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version 4.03
Overall survival | up to 5 years
  measured from first dose of iberdomide-cyclophosphamide-dexamethasone, to time of death from any cause. Patients still alive or lost to follow up are censored at the date they were last known to be alive.
Time to response | up to 5 years
  defined as time from first dose of iberdomide-cyclophosphamide-dexamethasone to the first objective documentation of PR or better.
Duration of response | up to 5 years
  defined as time from documentation of tumor response to disease progression.
Time to second objective disease progression (PFS2) | up to 5 years
  defined as time from first dose of iberdomide-cyclophosphamide-dexamethasone to 2nd disease progression or death from any cause.
Time to next treatment (TTNT) | up to 5 years
  defined as the date from first dose of iberdomide- cyclophosphamide-dexamethasone to first day when subject receives another myeloma treatment. Subjects who do not start new myeloma therapy are censored at the last known alive date or first dose date, whichever is later.

CONTACTS AND LOCATIONS:
Overall Officials: N.W.C.J van de Donk, Prof. MD PhD, Principal Investigator — Amsterdam UMC, location VUmc
Locations (9):
- Netherlands (9):
  - NWZ, Alkmaar
  - Amsterdam UMC, location AMC, Amsterdam
  - Amsterdam UMC, location VUmc, Amsterdam
  - Rijnstate, Arnhem
  - Amphia Ziekenhuis, Breda
  - Albert Schweitzer Ziekenhuis, Dordrecht
  - UMC Groningen, Groningen
  - Antonius ziekenhuis, Nieuwegein
  - Radboud UMC, Nijmegen

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Korst CLBM, Plattel W, de Kort EA, Smits F, Croockewit AJ, Levin MD, Westerman M, de Weerdt O, Nijhof IS, Wegman J, Smit N, Verkleij CPM, Mutis T, Nasserinejad K, Kerstiens R, van der Klift M, Franssen LE, de Ruijter MEM, Groen K, van der Spek E, Roeloffzen WWH, Zweegman S, van de Donk NWCJ. Iberdomide plus low-dose cyclophosphamide and dexamethasone in patients with relapsed and refractory multiple myeloma (the ICON study): a multicentre, single-arm, phase 2 trial. Lancet Haematol. 2026 Jan;13(1):e30-e40. doi: 10.1016/S2352-3026(25)00298-4. PMID 41482445